CLINICAL TRIAL: NCT02035124
Title: Cabazitaxel With BKM120 in Patients With Metastatic Castrate-Resistant Prostate Cancer Following Treatment With Docetaxel: Phase II Study With Safety Lead-in Cohort
Brief Title: Cabazitaxel and BKM120 in Patients With Metastatic Castrate-Resistant Prostate Cancer (mCRPC) Previously Treated With Docetaxel
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to slow accrual. No patients were enrolled.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 79
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Prostate Cancer
Keywords: Prostate; Metastatic; Refractory; mCRPC
MeSH Terms: conditions — Neoplasm Metastasis | interventions — NVP-BKM120; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 and Cabazitaxel (Experimental): BKM 120 orally once daily;
  Cabazitaxel 25 mg/m2 IV every 3 weeks
  Interventions: Drug: BKM 120; Drug: Cabazitaxel

INTERVENTIONS:
Drug: BKM 120
  Other Names: BKM 120 (Buparlisib)
Drug: Cabazitaxel
  Other Names: Jevtana

SUMMARY:
Although there have been advances in the treatment of patients with metastatic castrate-resistant prostate cancer (mCRPC), all patients eventually develop resistance to available therapy. Docetaxel is the accepted first-line agent followed by cabazitaxel in the post-docetaxel phase. In this study the investigators propose to evaluate BKM120, a PI3K inhibitor, with cabazitaxel in the treatment of patients with advanced prostate cancer.

DETAILED DESCRIPTION:
This study will be conducted in two parts. In a lead-in cohort, the feasibility and safety of administering BKM120 with a standard dose of cabazitaxel will be assessed. If safety is confirmed, a subsequent Phase II portion will assess the activity of the combination in patients with mCRPC previously treated with docetaxel. The treatment will consist of 3-week (21-day) cycles.

The ultimate purpose of this study will be to determine progression-free survival, response rate, disease control rate and overall survival of patients treated with the combination regimen and compare outcomes to historical results with single-agent cabazitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate confirmed histologically.
2. Metastatic disease confirmed by biopsy or imaging studies.
3. Patients must have received treatment with docetaxel as the only previous chemotherapy regimen. In addition, previous treatment with hormonal agents and/or immune therapy is allowed (e.g., abiraterone). (Previous treatment with MDV3100 will also be allowed.)
4. Patients must be castrate-resistant (i.e. developed progression of metastases following surgical castration or during medical androgen ablation therapy) with documented castrate levels of testosterone (<50 ng/dl).
5. Patients receiving medical castration therapy with gonadotropin-releasing hormone (GnRH) analogues should continue this treatment during this study.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2.
7. Patient must have progressive metastatic prostate cancer by at least 1 of the following criteria:

   * Soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
   * Bone scan progression defined by 2 or more new lesions on bone scan.
   * Prostate specific antigen (PSA) progression is determined by a minimum of three rising PSA levels with an interval of ≥1 week between each determination. The screening PSA measurement (documenting progression) must be ≥2 ng/mL.
8. Screening PSA ≥2 ng/mL.
9. Adequate hematologic, renal and hepatic function:
10. Adequate serum chemistries.
11. Ability to swallow and retain oral medication.
12. Life expectancy of ≥6 months.
13. Patients must be ≥18 years of age.
14. Patients entering this study must be willing to provide tissue from a previous tumor biopsy or 15 unstained slides (if available) for correlative testing. If tissue is not available, a patient will still be eligible for enrollment into the study.
15. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Previous treatment with PI3K inhibitors.
2. Known hypersensitivity to BKM120 or polysorbate-80 or any of the excipients or taxanes.
3. Use of an investigational drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of BKM120. For investigational drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the investigational drug and administration of BKM120 is required.
4. Previous chemotherapy with any agent other than docetaxel. All patients must be ≥28 days after their most recent chemotherapy and have recovered from side effects.
5. Patient has received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
6. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
7. Clinical significant peripheral neuropathy (defined as CTCAE v4.0 Grade ≥2) regardless of causality.
8. Mood disorders as judged by the Investigator or a Psychiatrist, or who meets the cut-off score of ≥12 in the Patient Health Questionnaire (PHQ)-9 or a cut-off score of ≥ 15 in the Generalized Anxiety Disorder (GAD)-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score or the PHQ-9)

   * anxiety or depression ≥ Grade 3
   * medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation, or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified
9. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if there is no evidence of central nervous system (CNS) disease progression, and at least 28 days (4 weeks) have elapsed since treatment. Patients are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs) during the study and should not be receiving chronic corticosteroid therapy for CNS metastases.
10. Leptomeningeal metastases or spinal cord compression due to disease.
11. Acute or chronic liver, renal disease or pancreatitis.
12. Uncontrolled diabetes mellitus. Type II diabetics are eligible if they require only oral hypoglycemic agents and fasting blood glucose level is ≤120. Type I diabetics are eligible if HbAlc is <8.
13. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, and malabsorption syndrome).
14. Any of the following cardiac diseases currently or within the last 6 months:

    * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
    * QTc > 480 ms on screening ECG
    * Unstable angina pectoris
    * Congestive heart failure (New York Heart Association [NYHA] ≥ Grade 2
    * Acute myocardial infarction
    * Conduction abnormality not controlled with pacemaker or medication
    * Significant ventricular or supraventricular arrhythmias (Patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible.)
    * Valvular disease with significant compromise in cardiac function.
15. Family history of congenital long or short QT, or known history of QT/QTc prolongation or Torsades de Pointes (TdP). Patients who are currently receiving treatment with medication that has the potential to prolong the QT interval or induce TdP and the treatment cannot either be discontinued or switched to a different medication prior to starting study treatment.
16. Inadequately controlled hypertension (i.e., SBP>180 mmHg or DBP>100mmHg). (Patients with values above these levels must have their BP controlled with medication prior to starting treatment)
17. Patient receiving chronic treatment with systemic steroids or another immunosuppressive agent at the start of study treatment.

    Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed.
18. Patients receiving drugs known to be moderate and strong inhibitors or inducers or isoenzyme cytochrome P450 (CYP) 3A (CYP3A) that cannot be discontinued or switched to different medication prior to starting study drug.
19. Patients who have taken herbal medications and certain fruits ≤7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
20. Patients currently receiving treatment with therapeutic doses of warfarin sodium. Patients receiving low molecular weight heparin are allowed.
21. A serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
22. Known diagnosis of human immunodeficiency virus (HIV), Hepatitis B (HBV) or Hepatitis C (HCV).
23. Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e. non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
24. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
25. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.
26. Fertile male patients, defined as all males physiologically capable of conceiving offspring must use a highly effective contraception during dosing any study agent + [5 x T1/2] +12 weeks = contraception through 16 weeks after final dosing of study therapy and should not father a child during this period. In addition, female partners of male patients must use a highly effective contraception during dosing of any study agent + [5 x T1/2] +12 weeks = contraception through 16 weeks after the final dose of study therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Serious and Non-Serious Adverse Events | up to 24 months
  Determine the optimal dose and safety of BKM120 given with cabazitaxel to patients with metastatic castrate-resistant prostate cancer.
Progression Free Survival (PFS) | every 6 weeks, up to 24 months
  time to disease progression

SECONDARY OUTCOMES:
Overall Response Rate | every 6 weeks, up to 24 months
  Percentage of complete responders (CR) or partial responders (PR) among patients evaluable for response
Overall Survival | up to 36 months
  Time from first treatment until death from any cause using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Tennessee Oncology PLLC, Nashville, Tennessee